CLINICAL TRIAL: NCT03090256
Title: Clinical Investigation of the AcrySof® IQ PanOptix™ IOL Model TFNT00
Brief Title: Clinical Investigation of the AcrySof® IQ PanOptix™ IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILH297-C003
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Cataract
Keywords: Trifocal IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PanOptix IOL (Experimental): AcrySof® IQ PanOptix™ IOL, bilateral implantation
  Interventions: Device: AcrySof® IQ PanOptix™ IOL

INTERVENTIONS:
Device: AcrySof® IQ PanOptix™ IOL — Multifocal intraocular lens (IOL) (near, intermediate, distance) implanted for long-term use over the lifetime of the cataract patient
  Other Names: Model TFNT00

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the AcrySof® IQ PanOptix™ Intraocular Lens (IOL) Model TFNT00 when implanted to replace the natural lens following cataract removal.

DETAILED DESCRIPTION:
Eligible subjects will attend a total of 10 visits over a 7-month period. Subjects will complete a preoperative examination of both eyes (Visit 0), followed by implantation of the IOL at the operative visit for each eye (Visit 00/00A), and up to 7 postoperative visits (each eye examined at Day 1-2 (Visit 1/1A), Day 7-14 (Visit 2/2A), and Day 30-60 (Visit 3/3A), with a binocular visit at Day 120-180 (Visit 4A) after the second implantation. The second implantation will occur within 30 days of the first.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign a statement of informed consent;
* Willing and able to complete all required postoperative visits;
* Cataracts in both eyes with planned cataract removal by phacoemulsification;
* Calculated lens power within the available range;
* Potential postoperative best corrected distance visual acuity (BCDVA) of 0.5 decimal or better in both eyes;
* Able to undergo second eye surgery within 30 days of the first eye surgery.

Exclusion Criteria:

* Significant irregular corneal aberration as demonstrated by corneal topography;
* Inflammation or edema (swelling) of the cornea affecting post-operative visual acuity;
* Degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted to cause future acuity losses;
* Previous refractive surgery;
* Diabetic retinopathy
* Other eye conditions as specified in the protocol
* Pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Group Manager, Clinical Development, Study Director — Alcon Japan, Ltd.
Locations (2):
- Japan (2):
  - Alcon Investigative Site, Fukuoka
  - Alcon Investigative Site, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 investigative sites located in Japan.
Pre-assignment Details: Of the 76 enrolled, 8 subjects were exited as screen failures prior to implantation. This reporting group includes all implanted subjects (68).
Groups:
- TFNT00: AcrySof® IQ PanOptix™ IOL, bilateral implantation
Period: Overall Study
Arm/Group | TFNT00
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all eyes with successful test article implantation (All-Implanted Analysis Set)
Arm/Group | TFNT00
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Monocular Photopic Best Corrected Distance Visual Acuity (5 m)
Description: Visual acuity (VA) was tested monocularly (each eye separately) under well-lit conditions with the subject's best spectacle correction at a distance of 5 meters (m) using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity. No hypothesis testing was planned for this study.
Time Frame: Visit 0 preoperative, Visit 1/1A (Day 1-2), Visit 2/2A (Day 7-14), Visit 3/3A (Day 30-60), Visit 4A (Day 120-180) post second implantation
Population: All-Implanted Analysis Set
Measure: Number; unit: subjects
Units Other Than Participants: Eyes
Groups:
- First Eye: AcrySof® IQ PanOptix™ IOL, first eye implantation
- Second Eye: AcrySof® IQ PanOptix™ IOL, second eye implantation
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 68 | 67
Number analyzed (Eyes) | 68 | 67
subjects
  Visit 0 preoperative: < 0.5 | 15 | 5
  Visit 0 preoperative: 0.5 - < 0.7 | 9 | 8
  Visit 0 preoperative: 0.7 - < 1.0 | 35 | 34
  Visit 0 preoperative: 1.0 or better | 9 | 20
  Visit 1/1A: < 0.5 | 0 | 0
  Visit 1/1A: 0.5 - < 0.7 | 1 | 0
  Visit 1/1A: 0.7 - < 1.0 | 8 | 8
  Visit 1/1A: 1.0 or better | 59 | 59
  Visit 2/2A: < 0.5 | 0 | 0
  Visit 2/2A: 0.5 - < 0.7 | 0 | 0
  Visit 2/2A: 0.7 - < 1.0 | 0 | 0
  Visit 2/2A: 1.0 or better | 68 | 67
  Visit 3/3A: < 0.5 | 0 | 0
  Visit 3/3A: 0.5 - < 0.7 | 0 | 0
  Visit 3/3A: 0.7 - < 1.0 | 2 | 1
  Visit 3/3A: 1.0 or better | 66 | 66
  Visit 4A: < 0.5 | 0 | 0
  Visit 4A: 0.5 - < 0.7 | 0 | 0
  Visit 4A: 0.7 - < 1.0 | 2 | 2
  Visit 4A: 1.0 or better | 66 | 65

2. Primary Outcome: Monocular Photopic Distance Corrected Intermediate Visual Acuity (60 cm)
Description: VA was tested monocularly under well-lit conditions using a chart. Distance-corrected VA at 60 cm is the VA at 60 cm measured under a corrected condition in which best-corrected VA at 5 m was obtained. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity. No hypothesis testing was planned for this study.
Time Frame: as for outcome 1
Population: All-Implanted Analysis Set
Measure: Number; unit: subjects
Units Other Than Participants: Eyes
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 68 | 67
Number analyzed (Eyes) | 68 | 67
subjects
  Visit 0 preoperative: < 0.5 | 47 | 40
  Visit 0 preoperative: 0.5 - < 0.7 | 18 | 18
  Visit 0 preoperative: 0.7 - < 1.0 | 1 | 8
  Visit 0 preoperative: 1.0 or better | 2 | 1
  Visit 1/1A: < 0.5 | 2 | 1
  Visit 1/1A: 0.5 - < 0.7 | 8 | 5
  Visit 1/1A: 0.7 - < 1.0 | 21 | 25
  Visit 1/1A: 1.0 or better | 37 | 36
  Visit 2/2A: < 0.5 | 0 | 0
  Visit 2/2A: 0.5 - < 0.7 | 1 | 0
  Visit 2/2A: 0.7 - < 1.0 | 13 | 7
  Visit 2/2A: 1.0 or better | 54 | 60
  Visit 3/3A: < 0.5 | 0 | 0
  Visit 3/3A: 0.5 - < 0.7 | 5 | 1
  Visit 3/3A: 0.7 - < 1.0 | 5 | 8
  Visit 3/3A: 1.0 or better | 58 | 58
  Visit 4A: < 0.5 | 2 | 1
  Visit 4A: 0.5 - < 0.7 | 3 | 3
  Visit 4A: 0.7 - < 1.0 | 4 | 7
  Visit 4A: 1.0 or better | 59 | 56

3. Primary Outcome: Monocular Photopic Distance Corrected Near Visual Acuity (40 cm)
Description: VA was tested monocularly under well-lit conditions using a chart. Distance-corrected VA at 40 cm is the VA at 40 cm measured under a corrected condition in which best-corrected VA at 5 m was obtained. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity. No hypothesis testing was planned for this study.
Time Frame: as for outcome 1
Population: All-Implanted Analysis Set
Measure: Number; unit: subjects
Units Other Than Participants: Eyes
Arm/Group | First Eye | Second Eye
Number analyzed (Participants) | 68 | 67
Number analyzed (Eyes) | 68 | 67
subjects
  Visit 0 preoperative: < 0.4 | 48 | 40
  Visit 0 preoperative: 0.4 or better | 20 | 27
  Visit 1/1A: < 0.4 | 1 | 0
  Visit 1/1A: 0.4 or better | 67 | 67
  Visit 2/2A: < 0.4 | 0 | 0
  Visit 2/2A: 0.4 or better | 68 | 67
  Visit 3/3A: < 0.4 | 0 | 0
  Visit 3/3A: 0.4 or better | 68 | 67
  Visit 4A: < 0.4 | 2 | 1
  Visit 4A: 0.4 or better | 66 | 66

ADVERSE EVENTS:
Time Frame: IOL implantation through study completion, an average of 6 months
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a subject, user, or other persons regardless of whether or not the event has a causal relationship with the medical device(s) or test procedure(s) in the study. Safety was assessed at each visit. This analysis population includes all eyes with attempted implantation (successful or aborted after contact with the eye) (Safety Analysis Set).
Groups:
- TFNT00: All subjects implanted with AcrySof® IQ PanOptix™ IOL
Arm/Group | TFNT00
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03090256/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT03090256/SAP_001.pdf